CLINICAL TRIAL: NCT07406789
Title: Phase II, Prospective, Randomized, Proof-of-Concept Study to Evaluate the Effects of a Personalized Dietary Intervention in Women With Advanced Gynecologic or Breast Tumors Treated With Antibody-Drug Conjugates (ADCs).
Acronym: LUMInova
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: TNC Nutrición Terapéutica S.L. (Other)
Collaborators: Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LMCA 001-2025 (LUMInova)
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Gynecologic Cancers; Advanced Breast Cancer
Keywords: Breast cancer; Diet; Cancer; Gynecologic
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (intervention) (Experimental): Personalised dietary intervention, tailored to clinical and metabolic parameters and individual preferences.
  Interventions: Dietary Supplement: Personalised dietary intervention.
- Cohort B (Control) (Active Comparator): General recommendations on the Mediterranean diet, without active dietary intervention.
  Interventions: Behavioral: General recommendations

INTERVENTIONS:
Dietary Supplement: Personalised dietary intervention. — Personalised dietary intervention, tailored to clinical and metabolic parameters and individual preferences.
  Other Names: Personalised diet
  Arms: Cohort A (intervention)
Behavioral: General recommendations — General recommendations on the Mediterranean diet, without active dietary intervention.
  Other Names: Mediterranean Diet
  Arms: Cohort B (Control)

SUMMARY:
The objective of the study is to evaluate the effect of a personalized dietary intervention (cohort A), compared with a standard nutritional intervention based on general recommendations for following a Mediterranean diet (cohort B), in women with advanced solid tumors of gynecologic or breast origin who are receiving treatment with antibody-drug conjugates (ADCs). This intervention is exclusively nutritional and does not involve the use of any investigational drug.

DETAILED DESCRIPTION:
Phase II, proof-of-concept, prospective, interventional, randomized, open-label study designed to evaluate the effect of a personalized dietary intervention on global quality of life in women with advanced gynecologic or breast tumors undergoing treatment with ADCs.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent to participate in the study, obtained prior to performing any specific procedure.
2. Women aged ≥ 18 years.
3. Confirmed diagnosis of advanced, incurable (stage IV or unresectable stage III) breast cancer or gynecologic cancer. This includes cancers of the breast, ovary, cervix, uterus, endometrium, fallopian tubes, vagina, or vulva.
4. Participants must have received a first cycle of ADC treatment in any line of treatment.
5. ECOG performance status 0-2.
6. Availability of their main clinical data with the possibility of follow-up.

Exclusion Criteria:

1. Male patient.
2. BMI <18 or > 40 kg/m2.
3. Patients with a life expectancy of less than 3 months.
4. Type 1 diabetes mellitus, metabolic diseases, and severe gastrointestinal disorders that interfere with the digestion or absorption of nutrients, as well as patients with severe renal or hepatic impairment.
5. Planned participation in treatment within a double-blind clinical trial.
6. History of previous or concomitant malignant disease of any other type that could affect compliance with the protocol or interpretation of results. Patients with curatively treated basal cell carcinoma of the skin or in situ cervical cancer are eligible for the study.
7. Presence of concurrent diseases or clinical conditions that, in the investigator's judgment, may significantly interfere with participation in the study, particularly those that limit the ability to adequately use the required digital tools (APP and wearable device). Patients will not be excluded due to common comorbidities if they retain adequate cognitive functioning and digital familiarity to comply with study procedures.
8. Carriers of therapeutic electronic devices: pacemakers, defibrillators, and cardiac resynchronization devices (due to potential interference caused by the wearable).
9. Patients who, in the investigator's judgment, do not possess sufficient digital capability to comply with the study procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Confirmed diagnosis of advanced, incurable (stage IV or unresectable stage III) breast cancer or gynecologic cancer. This includes cancers of the breast, ovary, cervix, uterus, endometrium, fallopian tubes, vagina, or vulva.
Enrollment: 100 (Estimated)
Dates: Start 2026-02-11 (Estimated); Primary Completion 2028-02-11 (Estimated); Study Completion 2028-02-11 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of a personalized dietary intervention on health-related quality of life (HRQoL), compared with general recommendations for a Mediterranean diet, in women with advanced gynecologic or breast tumors treated with ADCs. | 24 months
  Quality of life will be measured using the validated EORTC QLQ-C30 questionnaire, considering as the primary variable the percentage of patients experiencing clinically relevant improvement, defined as an increase of ≥10 points in the overall score from baseline.

SECONDARY OUTCOMES:
Evaluate changes in mental health and psychological well-being. | 24 months
  Assess changes in mental health and psychological well-being using the GHQ-28 questionnaire. The assessment variable will be the change from the baseline score in the total result and in each of the subscales (somatic symptoms, anxiety/insomnia, social dysfunction, and severe depression). Patients will be classified into those with emotional distress and those without, and the evolution of the distribution will be observed throughout the follow-up.
Evaluate perceived toxicity and treatment-related symptoms. | 24 months
  Evaluate perceived toxicity and treatment-related symptoms through the PRO-CTCAE v5.0 questionnaire, focusing on adverse events of special interest including fatigue, nausea and vomiting, diarrhea, peripheral neuropathy, conjunctivitis, blurred vision and dry eyes, neutropenia, rash, alopecia, anemia, and hand-foot syndrome.

OTHER OUTCOMES:
Assess progression-free survival in real life (rwPFS) | 24 months
  Defined as the time from randomisation to clinical progression (based on symptomatic or radiological criteria or change in treatment due to progression) or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario 12 Octubre, Madrid, Madrid, Spain